CLINICAL TRIAL: NCT00194909
Title: An Open Label, Dose Finding Trial of Viagra for the Treatment of Neuropathic Pain (in Diabetes Mellitus)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Thomas Brannagan, MD Associate Professor of Clinical Neurology, Weill Cornell Medical College
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1103-032
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2008-03-25 (Estimated); Status verified 2008-03

CONDITIONS: Diabetic Neuropathy
MeSH Terms: conditions — Diabetic Neuropathies | interventions — Sildenafil Citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: sildenafil (Viagra)

SUMMARY:
The purpose of this study is to study if sildenafil (Viagra) is effective in improving neuropathic pain. This will be an open label study at 3 doses of sildenafil (25 mg, 50 mg and 100 mg). If this study suggests efficacy, the information will be used to plan a placebo controlled, double-blind study in the future.

DETAILED DESCRIPTION:
Neuropathic pain is a common problem resulting from a diverse group of disorders including nerve injuries and neuropathies related to diabetes and other disorders. Pharmacologic agents are available such as gabapentin, which can successfully treat many patients. For many however there is inadequate treatment available, due to lack of efficacy and poor tolerability and the need for new pharmacologic agents is recognized.

We propose to study if sildenafil is effective in improving neuropathic pain, in patients with diabetes mellitus. Our primary outcome will be a reduction in the weekly average 11 point Likert pain scale (0 - no pain, 10 - worst possible pain) at 8 weeks. Secondary outcomes will include the Rand-36 quality of life scale, McGill visual analogue scale (VAS) and a sleep interference scale.

This will be an open label study at 3 doses of sildenafil (25 mg, 50 mg and 100 mg). Patients will begin at 25 mg at night for 1 week. If pain continues, the dose will be increased to 50 mg at night for 1 week. If pain continues the dose will be increased to 100 mg at night. Subjects will be on the medication for 8 weeks. If this study suggests efficacy, the information will be used to plan a placebo controlled, double-blind study in the future.

We propose to study if sildenafil is effective in improving neuropathic pain. Our primary outcome will be a reduction in the weekly average 11 point Likert pain scale (0 - no pain, 10 - worst possible pain) at 8 weeks. Secondary outcomes will include the Rand-36 quality of life scale, McGill visual analogue scale (VAS) and a sleep interference scale.

This will be an open label study at 3 doses of sildenafil (25 mg, 50 mg and 100 mg). Patients will begin at 25 mg at night for 1 week. If pain continues, the dose will be increased to 50 mg at night for 1 week. If pain continues the dose will be increased to 100 mg at night. Subjects will be on the medication for 8 weeks. If this study suggests efficacy, the information will be used to plan a placebo controlled, double-blind study in the future.

ELIGIBILITY:
Inclusion Criteria:

* Patients with signs and symptoms of a diabetic peripheral neuropathy as diagnosed by a neurologist with neuropathic pain will be included. The pain will have been present for at least 6 months. Patients may be on other medications for neuropathic pain such as anti-epileptic medications or tricyclic anti-depressants, however must be on a stable dose for 4 weeks prior to and during the study. Eligible patients must have a score of at least 40 on the VAS.

Exclusion Criteria:

* Previous adverse reaction to viagra
* Blood pressure < 90/50 or > 170/100
* unstable angina
* retinitis pigmentosa,
* myocardial infarction stroke or life-threatening arrhythmia within the last 6 months
* hemoglobulin A1c > 11
* HIV infection
* history of priapism
* hepatic or renal failure
* pregnancy
* current or past use of nitrates

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2004-08; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Our primary outcome will be a reduction in the weekly average 11 point Likert pain scale (0 - no pain, 10 - worst possible pain) at 8 weeks.

SECONDARY OUTCOMES:
Secondary outcomes will include the Rand-36 quality of life scale, McGill visual analogue scale (VAS) and a sleep interference scale.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas H Brannagan, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Peripheral Neuropathy Center - Weill Cornell Medical College, New York, New York, United States